CLINICAL TRIAL: NCT04093765
Title: Operational Evaluation of Mass Screening and Treatment Using Ultrasensitive Rapid Detection Tests to Reduce P. Falciparum Incidence in a Malaria Elimination Program in Eastern Kayin State, Myanmar
Brief Title: Mass Screening and Treatment for Reduction of Falciparum Malaria
Acronym: MSAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: MAL17011
Record Dates: First submitted 2019-09-02; First posted 2019-09-18 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2021-10

CONDITIONS: Plasmodium Falciparum Malaria
Keywords: Ultrasensitive Rapid Diagnostic Test; Mass Screening and Treatment; Greater Mekong Subregion; Malaria Elimination Task Force
MeSH Terms: conditions — Malaria, Falciparum | interventions — Antimalarials

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sustained high incidence villages (Experimental): Villages classified as high incidence, low probability of elimination (P. falciparum cumulative incidence >84 cases/1000/year, in spite of >1 year of functioning malaria post) will be eligible to be included in group 1. Villages in this group will be addressed by MSAT waves of 10-15 villages. Interventions will consist of 1 Ultrasensitive Rapid Diagnostic Test (URDT) and antimalarials drugs.
  Interventions: Diagnostic Test: Ultrasensitive Rapid Diagnostic Test (URDT); Drug: Antimalarials
- Seasonal focal transmission villages/locations (Experimental): This group will follow the NMCP case/and foci investigation guidelines, but use URDT instead of standard RDT for screening. MSAT group 2 locations will be cluster of houses, villages or clusters of villages selected based on the results of case or foci/outbreak investigation. Interventions will consist of 1 Ultrasensitive Rapid Diagnostic Test (URDT) and antimalarials drugs.
  * Village inclusion after case investigation
  * Village inclusion after outbreak investigation
  Interventions: Diagnostic Test: Ultrasensitive Rapid Diagnostic Test (URDT); Drug: Antimalarials

INTERVENTIONS:
Diagnostic Test: Ultrasensitive Rapid Diagnostic Test (URDT) — Investigation will consist in 1 URDT.
  For P. falciparum URDT positive:
  * collection of 3x1cm dried blood spots on filter paper
  * administration of a supervised antimalarial treatment course to individuals for which a P. falciparum will have been detected by URDT.
  Specifically in group 1, a population list will be collected in each village prior to MSAT campaign and all participants will undergo:
  * collection of a 200 µL-aliquot of capillary blood for each participant to the screening during the MSAT intervention.
  * 1 URDT + collection of a 200µL-aliquot of capillary blood for each participant to the follow-up survey at M12.
Drug: Antimalarials — A safe, recommended treatment of P. falciparum malaria will be administered to URDT positive individuals based on participant's characteristics:
  * The standard regimen for participants without known antimalarial allergy, not pregnant and not breastfeeding, will be a 3-day supervised weight-adjusted DP course and a single low dose PMQ. The single low dose PMQ will be administered on the first day.
  * Pregnant women and in their 2nd or 3rd trimester, and breastfeeding mothers, will receive a DP course but no PMQ.
  * Pregnant women in their first trimester will receive an oral course of quinine+clindamycin (7 days).
  * Individuals with known drug allergy to piperaquine will be treated with AL (+/- sld PMQ as per their pregnancy/breastfeeding status)
  * Specific/complex cases will be assessed by a medic and referred to a health facility for treatment if necessary.

SUMMARY:
In this project, the investigators aim at an operational research deployment of Ultrasensitive Rapid Diagnostic Test (URDT) -based Mass Screening and Treatment (MSAT) in the Malaria Elimination Task Force (METF) elimination program. This intervention will be tested in two types of setting. In group 1, MSAT will be used in a programmatic setting in order to decrease the reservoir of asymptomatic carriers in high incidence villages (following the same principles and objective as previously deployed MDA interventions). In group 2, the investigators take advantage of the lighter framework of MSAT to use it as a reactive intervention in order to respond to malaria outbreaks in low to intermediate incidence villages. The MSAT intervention will be preceded with community-level consent and community engagement (CE) activities. MSAT will be conducted over a period of approximately 1 week in each hamlet, village or group of villages, and will consist in administering a P. falciparum URDT to all individuals agreeing to participate. A limited subgroup (expected 5-25%) will be found positive and receive supervised treatment over 3 days for the standard regimen (DP to cure asexual stage infection + single low-dose primaquine to destroy gametocytes). After this intervention, the incidence of clinical falciparum episodes will be monitored by the village MP. In group 1, a comparison of the prevalence at baseline and 12 months after MSAT intervention will be performed through a second URDT survey, in addition to which both baseline and 12-month surveys will include the collection of a 200µL capillary blood sample for reference detection in the laboratory.

The intervention will be evaluated primarily on its ability to reduce yearly cumulative incidence of clinical falciparum malaria compared to year before intervention. Additional evaluations of the impact of MSAT will include: in group 1, comparison of asymptomatic infection prevalence; and in group 2, modifications of the shape of the incidence curve following intervention.

Funder: Wellcome Trust grant reference 106698/B/14/Z

DETAILED DESCRIPTION:
STUDY DESIGN

Stepped-wedge open-label, non-randomized, cluster intervention.

This study will be performed in clusters (hamlet (isolated group of household, village, or group of village). The intervention will be conducted in two types of clusters, both corresponding to locations where an excess of case was detected.

Group 1: Sustained high incidence clusters, characterized by a yearly cumulative incidence >84 cases/1000/year

Villages in group 1 will be attributed an intervention a given year based on the cumulative incidence over the previous 12 months (METF stratification January, including the last 2 transmission seasons). The order of intervention will be decided based on logistic constraints and highest incidence.

Group 2: Focal transmission clusters, corresponding to locations where an epidemic alert has been signalled and confirmed (see definition of thresholds).

Villages in group 2 will be attributed an intervention based on P. falciparum incidence in the previous 4 weeks. In near-0 transmission area, an intervention will be conducted in each likely source location of transmission of a locally acquired case. In the other areas (METF1+METF2), the intervention will be triggered when the incidence is above the pre-defined epidemic threshold.

In each cluster, all inhabitants will be invited to undergo an URDT test to identify their infection status, and will receive the appropriate treatment according to their characteristics. Information on village inhabitants absent during the MSAT activities will be obtained from village population lists provided by the village headman and from household member declarations. During the URDT screening, all individuals will receive a unique identifying number that will be used to record demographic data in the MSAT paper logbook and to label URDT and reference sample.

Before and after MSAT intervention, incidence of clinical malaria episodes will be recorded at the MP (1 or several) serving the cluster receiving the intervention. No individual data will be collected to link clinical case participation, infection status and incidence of clinical episodes.

Participants from group 1 clusters will be invited to participate in a prevalence survey during MSAT and 12 months after, in order to evaluate the impact of the MSAT campaign on the asymptomatic carriage prevalence. This will require collection of a 200µL sample during the MSAT campaign and a second round of URDT screening with the collection of a 200µL sample, 12 months after MSAT.

STUDY PARTICIPANTS

Populations of villages with high P. falciparum incidence located in Eastern Kayin State, Myanmar.

SUMMARY RESULTS

In 2018, two rounds of mass screening and treatment (MSAT) using ultrasensitive RDT (hsRDT) were conducted in 17 villages. The first round was carried out in 10 villages. Despite relatively high screening numbers with an average village screening coverage of 80.5% (min= 74.2%, max= 86%), equivalent to 1,364 people in total, only 1.1% of those screened were P. falciparum positive by hsRDT (ultrasensitive malaria RDT). In the second round of MSAT, 6 villages in underwent hsRDT screening. Screening numbers in this round were lower than in round 1 with an average of 70% (min= 47.1%, max= 90.8%) of villagers screened, or 1,104 people in total, however a higher positivity rate by hsRDT was detected with 5.38% of all tests returning a positive P. falciparum result.

In 2019, MSAT was conducted in 12 villages. This round had a high hsRDT screening coverage with an average coverage of 95% (min = 92%, max= 98%) in 12 villages, equivalent to 3,074 people. However, only 2.67% of hsRDTs returned a positive result for P. falciparum.

The primary intervention and outcome were completed in 31th Dec 2019. During the observation period post MSAT period in 2020. We have found the limited evidence for sustained impact of MSAT at low levels of P. falciparum detection in following post MSAT months by using hsRDT.

ELIGIBILITY:
Inclusion Criteria:

* All persons living in the village or cluster of villages will be eligible for MSAT intervention.
* Individuals living in smaller settlements (permanent or temporary) within walking distance of a selected intervention village will also be eligible.
* Large "work-related" settlements in the vicinity of a targeted village (military camps, logging camp, mining site) will be approached by the team to be included in the screening and treatment activity. They will be included in the analysis as a unit within a cluster of villages if all the study information can be collected (including follow-up survey for Group 1).

Exclusion Criteria:

* Individuals who do not provide informed consent for both URDT screening and treatment in case of positive result. Individuals will be given the possibility to refuse the collection of the 200µL reference sample or the DBS collection but participate to URDT screening and treatment.
* Children <1 year old
* Individuals with a documented Pf-positive malaria RDT who received treatment (AL+sld PMQ) during the previous 7 days.

NB: Individuals who were diagnosed infected with PF and received a treatment between 7 and 30 days before the intervention are still likely to be URDT positive due to the persistence of HRP2, and this will result in treatment of individuals who are likely uninfected. However, in a high prevalence area or in an outbreak context, previous infection signals exposure, and DP will provide a protection against a likely re-infection.

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 5542 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Adjusted incidence rate ratio before/after MSAT | 12 month

SECONDARY OUTCOMES:
Prevalence of P. falciparum infection measured in the village by URDT and by reference method (group 1) | 12 months
Change in the incidence dynamics over the transmission season (group 2) | 3 years
The percentage of participant among village resident tested by URDT. | 3 years
% of P. falciparum positive samples by reference method which were positive by URDT and treated; % of P. falciparum negative samples by reference method which were positive by URDT and treated (group 1) | 3 years

OTHER OUTCOMES:
Cumulative incidence of falciparum malaria episodes before and after MDA/MSAT; prevalence of falciparum infection before and after MDA/MSAT | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: francois Nosten, PhD, Principal Investigator — Shoklo Malaria Research Unit
Locations (1):
- Shoklo Malaria Research Unit, Mae Sot, Changwat Tak, Thailand

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-20): https://cdn.clinicaltrials.gov/large-docs/65/NCT04093765/Prot_SAP_002.pdf